CLINICAL TRIAL: NCT04428814
Title: A Phase 1, 2-Part, Randomized, Double-Blind, Parallel-Group, Single-Dose Study to Compare the Pharmacokinetics, Safety and Immunogenicity of Three Subcutaneous Injection Formulations of Ustekinumab in Healthy Male Subjects
Brief Title: Study to Compare PK and Safety of Subcutaneous Injection of Ustekinumab and CT-P43 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P43 1.1
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CT-P43 (Part 1) (Experimental): 45mg single dose administration
  Interventions: Biological: CT-P43
- EU-approved Stelara (Part 1) (Active Comparator): 45mg single dose administration
  Interventions: Biological: EU-approved Stelara
- CT-P43 (Part 2) (Experimental): 45mg single dose administration
  Interventions: Biological: CT-P43
- EU-approved Stelara (Part 2) (Active Comparator): 45mg single dose administration
  Interventions: Biological: EU-approved Stelara
- US-licensed Stelara (Part 2) (Active Comparator): 45mg single dose administration
  Interventions: Biological: US-licensed Stelara

INTERVENTIONS:
Biological: CT-P43 — 45mg single dose
  Arms: CT-P43 (Part 1); CT-P43 (Part 2)
Biological: EU-approved Stelara — 45mg single dose
  Arms: EU-approved Stelara (Part 1); EU-approved Stelara (Part 2)
Biological: US-licensed Stelara — 45mg single dose
  Arms: US-licensed Stelara (Part 2)

SUMMARY:
This study is a Phase 1, 2-Part, Randomized, Double-Blind, Parallel-Group, Single-Dose Study to Compare the Pharmacokinetics, Safety and Immunogenicity of Three Subcutaneous Injection Formulations of Ustekinumab (CT-P43, EU approved Stelara, and US licensed Stelara) in Healthy Male Subjects.

DETAILED DESCRIPTION:
CT-P43 is being developed as a proposed biosimilar of Stelara (ustekinumab). This study will be conducted in 2 parts. In Part 1, subjects will be enrolled and randomized in a 1:1 ratio to receive a single dose (45 mg) of either CT-P43 or EU-approved Stelara to collect preliminary safety data for CT-P43. In Part 2, subjects will be enrolled and randomized in a 1:1:1 ratio to receive a single dose (45 mg) of CT-P43, EU-approved Stelara, or US-licensed Stelara to demonstrate PK similarity. Each part will proceed independently, and subjects will be randomized to either Part 1 or Part 2 of the study subsequently. All subjects in Part 1 and Part 2 will undergo the same assessments. In each treatment arm in Part 1 and Part 2, all subjects will receive a study drug subcutaneously via PFS. The randomization to treatment assignment will be stratified by study center and body weight as measured at baseline to balance subject weight across treatment groups. Subjects will be confined to the study center until all required 24-hour post-dose assessments have been completed and will be discharged on Day 2. Subsequent visits will be carried out on an out-patient basis up to EOS.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects, between the ages of 18 and 55 years.
2. Subject with a BMI between 18.5 and 29.9 kg/m2. Weight between 60 to 100 kg.
3. Subject must agree to use medically acceptable methods of contraception consistent with local regulations during the course of the study and for 18 weeks after administration of the study drug.
4. Subject is informed and able to understand the full nature and purpose of the study, including possible risks and side effects, and is given ample time and opportunity to read and understand this information.

Exclusion Criteria:

1. Subject has a prohibited medical history and/or current condition.
2. Subject is planning to father a child or donate sperm within 18 weeks after the administration of the study drug (Day 1).
3. Subject previously received any biologic agents
4. In the opinion of the investigator, the subject is not eligible for the study participation for any reason.
5. Subject is vulnerable.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 271 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Demonstrate PK similarity | through study completion, up to day 127
  under the concentration-time curve from time zero to infinity (AUC0-inf) of CT-P43, EU-approved Stelara, and US-licensed Stelara
Demonstrate PK similarity | through study completion, up to day 127
  maximum serum concentration (Cmax) of CT-P43, EU-approved Stelara, and US-licensed Stelara

CONTACTS AND LOCATIONS:
Locations (2):
- New Zealand (2):
  - Auckland Clinical Studies Limited, Grafton, Auckland
  - Christchurch Clinical Studies Trust Limited, Christchurch, Canterbury